CLINICAL TRIAL: NCT05525273
Title: Neoadjuvant and Postoperative Treatment With Dabrafenib and Trametinib in BRAF Mutated Papillary Craniopharyngioma
Brief Title: Treatment of BRAF ( B-Rapidly Accelerated Fibrosarcoma) Mutated Papillary Craniopharyngioma
Acronym: Swecranio
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eva Marie Erfurth, MD, PhD (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Eva Marie Erfurth, MD, PhD, Professor, Skane University Hospital
Organization: Skane University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ver 1-21
Record Dates: First submitted 2022-04-20; First posted 2022-09-01 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Craniopharyngioma
Keywords: BRAF mutation; Dabrafenib; Trametinib; Neoadjuvant; Postoperative
MeSH Terms: conditions — Craniopharyngioma | interventions — dabrafenib; trametinib

STUDY DESIGN:
Intervention Model Description: Phase 1, single arm, open label, multicenter.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dabrafenib and trametinib (Experimental): Dabrafenib 75 mg twice daily and trametinib 2 mg once daily
  Interventions: Drug: Oral dabrafenib and trametinib

INTERVENTIONS:
Drug: Oral dabrafenib and trametinib — Neoadjuvant or postoperative treatment of patients with verified BRAF mutated papillary craniopharyngioma

SUMMARY:
Subjects with papillary craniopharyngioma harboring a BRAF mutation will be treated with a BRAF + MEK inhibitor (dabrafenib + trametinib) after informed consent. Study participants will be administered oral dabrafenib and trametinib until maximal tumor volume reduction assessed by MRI. Progression free survival, cognition, ophthalmologic status, hypothalamic status and quality of life will be assessed 1 year after initiation of study treatment

DETAILED DESCRIPTION:
Background. Papillary craniopharyngioma harbours a BRAF mutation in 90% of cases. Treatment with BRAF + MEK (mitogen activated protein kinase ) inhibitors (dabrafenib + trametinib) may prevent patients from undergoing surgery with a high risk of serious side effects, or provide an additional treatment option when further surgery is not advised.

Study intervention Subjects with newly diagnosed craniopharyngioma where radical surgery is not considered adequate or patients with recurrence of craniopharyngioma where further surgery is not considered possible without serious sequelae will be asked for informed consent Study participants are treated continuously with dabrafenib and trametinib orally, until maximal tumor shrinkage. Evaluation is done by MRI to measure tumor volume, as well as assessment of performance status, quality of life, cognition, ophthalmologic status, performance status and hypothalamic status.

Study type The study is a Phase II, single armed, open label and multicenter study Study drugs are Dabrafenib (Tafinlar) and trametinib (Mekinist) Primary outcome To evaluate tumor response in the form of reduced tumor volume on MRI in patients with papillary craniopharyngioma during treatment with dabrafenib and trametinib.

Secondary outcomes

To evaluate dabrafenib and trametinib treatment for the following aspects:

* response according to RECIST Duration of response for patients treated without subsequent surgery
* how many patients become operable after neoadjuvant treatment
* progression-free survival after 1 and 2 years
* quality of life during and after treatment The effect of treatment on vision, cognition and hypothalamic effects Exploratory outcomes Levels of circulating BRAF Trial population 25 patients Trial duration Participants are treated with the study treatment for at least one year if the treatment is well tolerated, to maximum tumor reduction, or longer according to the investigators´s assessment. Treatment is discontinued in case of progression, unacceptable toxicity or at the request of the patient.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically verified papillary craniopharyngioma.
2. BRAF mutated V600E (valine 600 glutamine), verified immunohistochemically and by molecular genetic analysis
3. Newly diagnosed tumor, or recurrence after previous surgery, where surgery is not considered to be able to be performed radically without the risk of serious or permanent sequelae.
4. Age over 18 years
5. Functional status according to ECOG (Eastern Cooperative Oncology Group performance status) 0-2
6. Adequate organ function:

   neutrophils> 1.5 x 109 platelets> 100 x 109 creatinine <1.5 x ULN (upper limit of normal) or creatinine clearance <45 ml / min bilirubin <1.5 x ULN ASAT (aspartate aminotransferase) / ALAT (alanine aminotransferase) <2.5 x ULN
7. Ability to understand and give informed consent.
8. Previous cancer, which does not require current treatment is allowed.
9. The patient agrees to use an adequate method to avoid pregnancy.

Exclusion Criteria:

1. Ongoing treatment in another drug study or other experimental treatment.
2. Previous treatment with BRAF or MEK inhibitors.
3. Hypersensitivity to study drugs.
4. Ongoing treatment with non-authorized drugs, (strong inducers of CYP2C8 or CYP3A4). If the patient is on unauthorized drugs, they must be discontinued at least 14 days before inclusion.
5. Known cardiovascular disease where treatment with MEK inhibitors is considered inappropriate, eg severe heart failure, prolongation of QT time, uncontrolled arrhythmia, recent (<6 months) cardiac infarction, uncontrolled hypertension.
6. Active bleeding; intracranial hemorrhage last 4 weeks before inclusion.
7. Thromboembolic disease last 6 months and unstable anticoagulant treatment less than 4 weeks before inclusion.
8. Women who are pregnant or breastfeeding.
9. Previous central serous retinopathy or retinal vein occlusion.
10. Previous uveitis or iritis last 4 weeks before inclusion.
11. Surgery within the last 3 weeks.
12. For postoperative patients; radiation therapy within the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2027-09-10 (Estimated); Study Completion 2028-04-10 (Estimated)

PRIMARY OUTCOMES:
Tumor response | 1 month to 5 years (sliding timepoints)
  To evaluate tumor response measured as maximally reduced tumor volume on MRI during treatment with dabrafenib and trametinib. Maximally reduced volume is defined as the time point where no further reduction of tumor volume can be observed

SECONDARY OUTCOMES:
Response ratio | 1 year after initiation of study treatment
  Response ratio according to RECIST
Response duration | From time of study drug discontinuation to time of observed increased tumor volume assessed up to 1 year
  Duration of response for patients treated without subsequent surgery
Operability after neoadjuvant trial treatment | 1 year after initiation of study treatment
  Number of patients which become operable after neoadjuvant treatment
Progression-free survival 1 year | 1 year
  Defined as unchanged or diminished tumor volume
Progression-free survival 2 years | 2 years
  Defined as unchanged or diminished tumor volume
QOL after treatment | 1 year
  Quality of life assessed by EQ5D5L (EuroQual 5 dimensions 5 levels) at 1 year after start of study treatment and compared to baseline
QOL after treatment | 1 year
  Quality of life assessed by EORTC QLQ30 (European Organisation for Research and Treatment of Cancer-Quality of Life Questionnaire 30) at 1 year after start of study treatment and compared to baseline
Cognitive status after treatment | 1 year
  Cognitive status assessed by CNS (central nervous system) Vital Signs 1 year after initiation of treatment and compared to baseline
Opthalmologic status after treatment | 1 year
  Opthalmologic status assessed as compound measure of visual acuity and visual field defects 1 year after initiation of treatment and compared to baseline
Hypothalamic status after treatment | 1 year
  Hypothalamic status assessed as compound measure of pituitary and hypothalamic status 1 year after initiation of treatment and compared to baseline

OTHER OUTCOMES:
Levels of circulating mutated BRAF | 1 week after initiation of trial treatment
  BRAF assessed by plasma analysis and compared to baseline levels
Levels of circulating mutated BRAF | 2 weeks after initiation of trial treatment
  BRAF assessed by plasma analysis and compared to baseline levels
Levels of circulating mutated BRAF | 6 months after initiation trial treatment
  BRAF assessed by plasma analysis and compared to baseline levels
Levels of circulating mutated BRAF | 12 months after initiation trial treatment
  BRAF assessed by plasma analysis and compared to baseline levels
Levels of circulating of mutated BRAF | 3 months after end of trial treatment
  BRAF assessed by plasma analysis and compared to baseline levels

CONTACTS AND LOCATIONS:
Overall Officials: Peter Siesjö, MD. PhD., Study Chair — Department of Neurosurgery, SUS, Lund Sweden; Sara Kinhult, MD. PhD, Study Chair — Department of Oncology, SUS, Lund Sweden; Eva Marie Erfurth, MD. PhD, Principal Investigator — Department of Endocrinology, SUS, Lund, Sweden
Locations (1):
- Department of Endocrinology, Lund, Sweden